CLINICAL TRIAL: NCT06659965
Title: Intravenous Methocarbamol for Acute Pain After Spine Surgery
Acronym: IMAPSS
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Paul Potnuru, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-24-1095; 5T32GM135118-03 (NIH)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Acute Post Operative Pain; Postsurgical Pain Management; Spine Surgery; Acute Pain, Postoperative; Multimodal Analgesia
Keywords: methocarbamol; postoperative pain; Robaxin; spine surgery; acute postsurgical pain; postsurgical pain; target trial emulation; postoperative analgesia; postoperative pain management; multimodal pain management
MeSH Terms: conditions — Pain, Postoperative | interventions — Methocarbamol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IV methocarbamol: Patients who received intravenous methocarbamol
  Interventions: Drug: Intravenous Methocarbamol
- Usual Care: Patients who received usual postoperative pain management after surgery without any intravenous methocarbamol administration

INTERVENTIONS:
Drug: Intravenous Methocarbamol — At least 500 mg of intravenous methocarbamol administered within 2 hours after the end of elective spine surgery for acute postoperative pain management
  Other Names: Robaxin
  Groups: IV methocarbamol

SUMMARY:
The goal of this target trial emulation is to evaluate the impact of intravenous (IV) methocarbamol on postoperative pain and opioid use in adults undergoing elective spine surgery. The main questions it aims to answer are:

* Does IV methocarbamol reduce pain in the 6 hours following surgery?
* Does IV methocarbamol decrease the need for opioid pain medications in the same period?

Participants who receive IV methocarbamol as part of their routine postoperative care will have their pain scores and opioid consumption tracked for 6 hours after treatment. Pain levels will be measured using standard assessments, and opioid use will be quantified in oral morphine equivalents.

DETAILED DESCRIPTION:
The IMAPSS study is a target trial emulation evaluating the effect of intravenous (IV) methocarbamol on postoperative pain management and opioid consumption in adult patients undergoing elective spine surgery. The study employs a target trial emulation design to simulate the conditions of a randomized controlled trial using observational data extracted from electronic medical records. The main focus is to determine if administering IV methocarbamol within two hours after surgery reduces postoperative pain scores and opioid use.

Patients will be tracked from the point of their first recorded pain score in the Post-Anesthesia Care Unit (PACU) after surgery to assess for treatment assignment eligibility. Data will be collected at 15-minute intervals, which corresponds to the standard assessment frequency in Phase I PACU care, for up to 12 hours postoperatively for each patient. The primary analysis will use time-varying propensity score matching (TV-PSM) to control for baseline and time-varying confounders. Pain levels will be measured using a time-weighted average (TWA) of pain scores, and opioid consumption will be quantified in oral morphine equivalents (OME).

The primary analysis will utilize TV-PSM, with propensity scores estimated through a Cox proportional hazards model. Matching will create balanced treatment groups at each 15-minute interval. Generalized estimating equations (GEE) will then estimate the effect of IV methocarbamol on the primary outcome (TWA pain) and secondary outcome (cumulative OME) over a 6-hour postoperative period. As a sensitivity analysis, a marginal structural model (MSM) using inverse probability weighting (IPW) will assess the robustness of the findings to the time-varying confounder adjustment.

This study's findings will aim to inform evidence-based recommendations for postoperative pain management and opioid-sparing strategies, potentially providing safer alternatives to conventional opioid-based regimens.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing one of the following three elective spine surgeries: (i) Anterior Cervical Discectomy and Fusion (ACDF), (ii) Posterior Spinal Fusion, or (iii) Laminectomy, Laminotomy, or Discectomy
* At least 8h of valid pain scores recorded postoperatively

Exclusion Criteria:

* Emergency Surgery
* Pregnancy
* Sensitivity to methocarbamol (allergy)
* End-stage renal disease (ESRD)
* Myasthenia gravis
* Missing a valid electronic anesthesia record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing elective spine surgeries at multiple hospitals within a large health system in Houston, TX. This includes individuals receiving surgical interventions for conditions such as degenerative disc disease, spinal stenosis, or other spinal pathologies that require procedures like ACDF, posterior spinal fusion, or laminectomy. Participants will be selected from those who receive perioperative care across various hospital settings within the health system, including postoperative management in the Post-Anesthesia Care Unit (PACU).
Sampling Method: Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Time-Weighted Average Pain Score | 6 hours after treatment assignment
  The primary outcome of this study is the Time-Weighted Average (TWA) pain score measured over the 6-hour period following treatment assignment. Pain scores are collected using a standardized numerical pain rating scale, ranging from 0 (no pain) to 10 (worst possible pain). These scores are assessed in 15-minute intervals, the standard frequency for Phase I PACU assessments, throughout the 6-hour follow-up period. The TWA pain score is calculated by averaging these pain ratings, giving greater weight to scores recorded more frequently or for longer periods. This method provides a comprehensive summary of the patient's pain experience over the observed time frame, accounting for fluctuations in pain intensity during recovery. A lower TWA score indicates better pain control and a potentially greater effect of the intervention.

SECONDARY OUTCOMES:
Cumulative Opioid Use | 6 hours after treatment assignment
  The secondary outcome of this study is the cumulative opioid use measured in Oral Morphine Equivalents (OME) over the 6-hour period following treatment assignment. Opioid doses administered during this timeframe are converted into OME to standardize and compare the total amount of opioids used, accounting for the specific medication, dose, and route of administration. Data on opioid administration are assessed in 15-minute intervals, aligned with standard PACU assessment practices. The cumulative OME reflects the total opioid exposure a patient received, providing a quantitative measure of opioid consumption and its potential reduction with the intervention. Lower cumulative OME values suggest more effective pain management with fewer opioids, indicating the potential benefits of non-opioid alternatives.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Potnuru, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Health System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) used in the publication of the results will be shared with interested researchers upon request when the required documentation is completed, and a review by the study team is completed and approved.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2025-January 2027
Access Criteria: A proposal that describes planned analyses must be submitted by email to the corresponding author. The study team will review the request before approval.

REFERENCES:
- [Background] Potnuru P, Baranov A, Khudirat M, Turan A. Intravenous methocarbamol for acute pain after spine surgery: a target trial emulation. Reg Anesth Pain Med. 2025 Sep 8:rapm-2025-107010. doi: 10.1136/rapm-2025-107010. Online ahead of print. PMID 40921494